CLINICAL TRIAL: NCT06530888
Title: Feasibility of Process-based Therapy in a Naturalistic Setting
Acronym: PBaPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ulrich Stangier, Director of the Department of Clinical Psychology and Psychotherapy and Center for Psychotherapy, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: III L5 - 519/05.000.002 - 2
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Depressive Disorder; Anxiety Disorder
Keywords: feasibility; Process-based Therapy
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Process-based Cognitive Behavioral Therapy (Experimental): In PBT, treatment planning is based on a dynamic network analysis of EMA data collected during the baseline phase. Therapists identify the central node, significant edges, self-loops, and feedback loops between the nodes. Using this information, interventions are selected based on empirical evidence for mechanisms of change that correspond to the network characteristics.
  These interventions are framed within an evolutionary framework as the variation, selection, and retention of an adaptive mode of the central node in relation to the specific context of the problem. The change in this key variable is monitored through daily judgments based on EMA. Treatment also focuses on additional targets to establish adaptive modes of the dimensions as defined in the positive network model. Concomitant medication is allowed and will be controlled in statistical analyses.
  Interventions: Other: Process-based Cognitive Behavioral Therapy (PBT)
- Routine practice (r-PT) (Active Comparator): In r-PT, as opposed to PBT, a naturalistic setting is retained for treatment decisions. Treatment planning follows traditional theories about the factors maintaining the disorder and interventions changing them, e.g. avoidance and exposure in anxiety disorders or reduced reinforcement of activities and behavioral activation in depression. Interventions are based on common treatment manuals related to diagnoses, e.g. CBT for depression. Individual data from the behavioral analysis are used to tailor the techniques to the individual problems of the patients. Treatment process is largely structured by personal preferences of the therapist due to experience, knowledge or recommendations of the National guidelines for the mental health problem.Concomitant medication is allowed and will be controlled in statistical analyses.
  Interventions: Other: Routine practice (r-PT)

INTERVENTIONS:
Other: Process-based Cognitive Behavioral Therapy (PBT) — Intervention planning based on the use of EMA data, feedback of dynamic network analysis and matching of interventions to central nodes of the network.
  Other Names: Process-based Therapy with Ecological Momentary Assessment
  Arms: Process-based Cognitive Behavioral Therapy
Other: Routine practice (r-PT) — Intervention planning as usual.
  Arms: Routine practice (r-PT)

SUMMARY:
The main objective is to explore the feasibility of Process-based Therapy in a natural mental health care setting delivered by practitioners.

DETAILED DESCRIPTION:
In the naturalistic setting of mental health care, treatment decisions of psychotherapists are often based on theories or experience related to treatment approaches. An alternative approach to treatment decision is suggested by Process-based Therapy (PBT), which emphasizes empirical and rational criteria for the selection of intervention. It utilizes ecological momentary assessment (EMA) data, incorporates feedback from dynamic network analysis, and supports interventions based on individual network models and empirical evidence from research related to change processes. Currently, there are no data on the feasibility and acceptability of PBT in practice. The present study investigates in a naturalistic setting, whether PBT can be implemented by psychotherapists in mental health care. Furthermore, the investigators explore the acceptability and efficacy of PBT as compared to psychotherapy delivered in routine practice (r-PT).

ELIGIBILITY:
Inclusion Criteria:

* A primary DSM-5 diagnosis of a depressive or anxiety disorder
* Age 18-65 years
* Sufficient knowledge of the German language
* Participating patients are not required to discontinue medication, but to keep medication constant over the treatment period

Exclusion Criteria:

* Increased suicidality
* Substance abuse or dependency
* Diagnose of a cluster A or B (DSM-5) personality disorder
* Pervasive developmental disorder
* Psychotic disorder
* Eating disorder
* Bipolar disorder
* Severe physical illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Credibility/expectancy questionnaire(CEQ) | Assessed at pre-treatment
  Treatment expectancy and credibility, minimum value= 4, maximum value= 56, higher scores mean better outcome
Patient attitude towards utility of EMA and networks Scale (PAUEN) | Assessed at post-treatment (week 28)
  Attitude towards utility of EMA and network models, minimum value= 8, maximum value= 40, higher scores mean better outcome
Therapist attitude towards utility of EMA and networks Scale (TAUEN) | Assessed at post-treatment (week 28)
  Attitude towards utility of EMA and network models, minimum value= 6, maximum value= 30, higher scores mean better outcome
Treatment Evaluation Inventory (TEI) | Assessed at post-treatment (week 28)
  Acceptance of treatment, minimum value= 7, maximum value= 98, higher scores mean better outcome

SECONDARY OUTCOMES:
Euroqol-5D (EQ-5D) | Assessed at pre-treatment, at post-treatment (week 28) and at 6-month follow-up
  Health related quality of life, minimum health state=11111, maximum health state=55555, higher scores in health state mean worse outcome, minimum health score=0, maximum health score=100, higher scores in health score mean better outcome
Positive-Mental Health Scale (PMH) | Assessed at pre-treatment, at post-treatment (week 28) and at 6-month follow-up
  Psychological wellbeing, minimum value=9, maximum value=36, higher scores mean better outcome
Depression Anxiety Stress Scale (DASS-10) | Assessed at pre-treatment, at intermediate treatment (week 8), at post-treatment (week 28) and at 6-month follow-up
  Psychological symptoms of distress, depressive and anxious symptoms, minimum value=0, maximum value=30, higher scores mean worse outcome
Acceptance and Action Questionnaire Version 2 (AAQ-2) | Assessed at pre-treatment, at intermediate treatment (week 8), at post-treatment (week 28) and at 6-month follow-up
  Psychological flexibility and acceptance, minimum value=7, maximum value=49, higher scores mean worse outcome
Reflective Functioning Questionnaire (RFQ-8) | Assessed at pre-treatment, at intermediate treatment (week 8), at post-treatment (week 28) and at 6-month follow-up
  Reflective Functioning, minimum value=8, maximum value=56, higher scores on the uncertainty dimension mean worse outcome, higher scores in the certainty dimension mean better outcome
Process-based Assessment Tool (PBAT) | Assessed at pre-treatment, at intermediate treatment (week 8), at post-treatment (week 28) and at 6-month follow-up
  Variation, selection and retention of adaptive behavior, minimum value=0, maximum value=1800, higher scores mean better outcome
Cognitive-Behavioral-Therapy Skills Questionnaire (CBTSQ) | Assessed at pre-treatment, at intermediate treatment (week 8), at post-treatment (week 28) and at 6-month follow-up
  Patients use of CBT interventions, minimum value=6, maximum value=42, higher scores mean better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- JWGUniversity, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the main publication of outcomes, after deidentification (text, tables, figures, and appendices) will be shared. Further Study Protocol, Analysis Plan, Informed Consent Form and Analytic Code will be shared to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication. Data are available for 5 years at a third-party website (Link to be included).
Access Criteria: Proposals should be directed to stangier@psych.uni-frankfurt.de. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- See also: University website — https://www.psychologie.uni-frankfurt.de/140318315/PBaPP_Patienteninformation

DOCUMENTS (1):
  • Study Protocol (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT06530888/Prot_000.pdf